CLINICAL TRIAL: NCT01952470
Title: Investigating the Role of Nebulised Mucolytic Therapy During Lower Respiratory Tract Infections Post Lung Transplantation.
Brief Title: Preliminary Study of Dornase Alfa to Treat Chest Infections Post Lung Transplant.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: The Alfred Research Trusts Small Project Grant. (Unknown); Dr Carey Denholm and Laura Denholm (Unknown)
Responsible Party: Principal Investigator, Benjamin Tarrant, Benjamin James Tarrant, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 342/13; DOI:10.1111/tri.13400 (Other: Transplant International - journal)
Record Dates: First submitted 2013-08-31; First posted 2013-09-30 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Lung Transplant Infection; Lower Respiratory Tract Infection
Keywords: Lung transplantation; Respiratory Tract Infections; Respiratory Therapy; Isotonic Solutions; Sodium Chloride; Postoperative complications; Postoperative care; dornase alfa
MeSH Terms: conditions — Respiratory Tract Infections; Postoperative Complications | interventions — dornase alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dornase Alfa (Experimental): Once daily, 2.5ml inhaled dornase alfa.
  Interventions: Drug: Dornase Alfa
- Isotonic Saline (Active Comparator): Once daily, 5ml inhaled 0.9% normal saline.
  Interventions: Drug: Isotonic Saline.

INTERVENTIONS:
Drug: Dornase Alfa — Once daily, 2.5ml inhaled dornase alfa (evening if able) with inhalational breathing routine (IBR). IBR consists of 4 slow deep breaths followed by 6 relaxed breaths, repeated until nebuliser is complete, coughing when the patient feels the need to expectorate. The patient will be instructed to sit in an upright position with upper limb support as able.
  Other Names: Pulmozyme.
  Arms: Dornase Alfa
Drug: Isotonic Saline. — Once daily, 5ml inhaled 0.9% normal saline (evening if able) with inhalational breathing routine (IBR). IBR consists of 4 slow deep breaths followed by 6 relaxed breaths, repeated until nebuliser is complete, coughing when the patient feels the need to expectorate. The patient will be instructed to sit in an upright position with upper limb support as able.
  Other Names: normal, 0.9% saline.
  Arms: Isotonic Saline

SUMMARY:
Patients who have undergone lung transplantation are at an increased risk of developing chest infections due to long-term medication suppressing the immune response. In other chronic lung diseases such as cystic fibrosis (CF) and bronchiectasis, inhaled, nebulised mucolytic medication such as dornase alfa and isotonic saline are often used as part of the management of lung disease characterized by increased or retained secretions. These agents act by making it easier to clear airway secretions, and are currently being used on a case-by-case basis post lung transplantation.

To the investigators knowledge, these agents have not been evaluated via robust scientific investigation when used post lung transplant, yet are widely used in routine practice. Patients post lung transplant must be investigated separately as they exhibit differences in physiology that make the clearance of sputum potentially more difficult when compared to other lung diseases. Lower respiratory tract infections are a leading cause of hospital re-admission post lung transplant. Therefore, this highlights the need for a randomized controlled trial. The aim of this study is to assess the efficacy of dornase alfa, compared to isotonic saline, in the management of lower respiratory tract infections post lung transplant. Investigators hypothesize that dornase alfa will be more effective than isotonic saline.

The effect of a daily dose of dornase alfa and isotonic saline will be compared over a treatment period of 1 month. Patients admitted to hospital suffering from chest infections characterized by sputum production post lung transplant will be eligible for study inclusion. Patients will be followed up through to 3 months in total to analyze short-medium term lasting effect. Investigators wish to monitor physiological change within the lung non-invasively via lung function analysis whilst assessing patient perceived benefit via cough specific quality of life questionnaires. These measures will be taken at study inclusion and repeated after 1 month and 3 months. Day to day monitoring will be performed via patient symptom diaries, incorporating hospital length of stay and exacerbation rate. The outcomes of this study have the potential to guide clinical decision-making and highlight safe and efficacious therapies.

DETAILED DESCRIPTION:
According to the International Society for Heart and Lung Transplantation (ISHLT), the incidence of lung transplants per annum worldwide is rising annually, with over 3000 transplants completed according to the latest registry(1). The Alfred is a state-wide, internationally renowned lung transplant service, transplanting between 59 - 79 patients over the last two calendar years, with a wait-list of more than 40 potential recipients. This makes it one of only 7 centres worldwide completing this volume of transplants(1).

Patients who have undergone lung transplantation for end-stage lung disease are subject to life-long immunosuppression to prevent allograft rejection. These patients are at a heightened risk of acquiring opportunistic lower respiratory tract infections (LRTI)(2), often characterized by sputum retention and / or production, which can have a negative impact on both morbidity and mortality(3). Patients post lung transplant often find it difficult to clear secretions due to an alteration in normal physiology. Transplanted lung tissue is denervated upon resection from the donor, which has been shown to lead to slower cilial beat frequencies(4), impaired muco-ciliary clearance (MCC) rates(4-6) and an impaired cough reflex(7). Devascularisation to lung tissue post ischaemic surgical time in the acute period can lead to an alteration in mucosal properties and structural changes around anastomoses, which may further impair the ability to clear secretions(3).

Inhaled, nebulised mucolytic agents are commonly used in the management of other suppurative chronic lung diseases characterized by excessive production of secretions. Dornase alfa acts by digesting the extracellular deoxyribonucleic acid (DNA) released by inflammatory cells during infection(8). It has been shown to have positive long-term effects on lung function in cystic fibrosis (CF)(8) and short-term benefits treating atelectasis and mucous plugging in acute, non-CF adult and pediatric cases(9-11). Yet shown to be safe in normal subjects(8), it has been shown to have a detrimental effect on pulmonary function in non-CF bronchiectasis(12).

Inhaled saline acts by restoring the airway surface liquid layer of the mucosa, favorably altering mucous properties, accelerating MCC and stimulating cough(13-14). Positive evidence exists for hypertonic saline (6-7%) in CF(13-14) and both hypertonic and isotonic (0.9%) saline in non-CF bronchiectasis(15). There is discussion of clinical use of saline as a mucolytic in the post transplant patient(16) with no evidence by way of randomized controlled trial to demonstrate effect. There is no current evidence on the use of inhaled mucolytics post transplant.

Currently, both dornase alfa and saline (isotonic / hypertonic) are used in the inpatient and outpatient setting at this institution as a reactive treatment strategy for LRTI characterized by excessive sputum production and / or retention. The investigators believe this warrants a short-term, randomized trial to assess the efficacy of current practice, and to evaluate whether dornase alfa is more effective than 0.9% saline, a cheaper, more accessible alternative.

Aim

To evaluate the efficacy of inhaled dornase alfa compared to inhaled isotonic (0.9%) saline on:

* Quantitative and qualitative respiratory outcomes
* The need for antibiotics, length of stay and exacerbation / re-admission rates

Hypothesis Dornase alfa is more effective than isotonic saline in the post lung transplant population during LRTI.

Study design Phase 2, assessor blinded, prospective randomized controlled trial.

Intervention On admission to the ward as an inpatient, patients who give informed consent within 48 hours of initial presentation will be randomly assigned to one of two groups defined below. The randomization sequence will be concealed using opaque envelopes. Randomization will be stratified according to pre-transplant diagnosis (cystic fibrosis or not) as people with cystic fibrosis are expected to be younger and have a different underlying systemic disease process.

All participants will undertake treatment for one month according to their allocated group, with follow up to 3 months, (2 months off randomized intervention). Both groups will continue to do their regular prescribed physical exercise routine over the course of the study.

Timing of assessment All outcome measures will be performed at study baseline, 1 month and 3 months follow-up. Daily outcome measures used as a monitoring diary are an exception. There are no cough-specific quality of life questionnaires validated for use in the post lung transplant population.

Sample size and power calculation A total of 30 participants (15 in each group) will enter this study. The probability is 80 percent that the study will detect a treatment difference at a two-sided 0.05 significance level, if the true difference between treatments is 1.000 unit in lung clearance index (LCI).

This is a conservative estimate that is smaller than previous differences found in pediatric populations(17-18). This is based on the assumption that the standard deviation of the response variable is 0.94 units(17-18).

As a phase 2 study, this project is powered to detect differences in physiological outcomes, rather than quality of life or hospitalization. However, should the treatment prove to have physiological benefits, the secondary outcomes of this study will provide critical information for powering a future phase 3 trial.

Feasibility: Approximately 12 patients with pulmonary exacerbations are admitted under the lung transplant service each month (minimum estimate). Investigators estimate that 70% will meet the eligibility criteria for the study and 50% will consent to participate. It is therefore anticipated that it will be possible to recruit the numbers needed for this study in 8 months.

Statistical analysis An intention to treat analysis will be conducted, with inclusion of all randomized participants, regardless of study completion. Data for continuous outcomes including LCI will be analyzed using a linear mixed models analysis, which makes use of all available data at each time point and is less affected by incomplete data than analysis of variance. The likelihood of exacerbation or hospitalization during the follow-up period for the dornase alpha group will be expressed as a relative risk compared to the isotonic saline group.

Bias / Confounders There is potential for performance bias in this study due to the lack of ability to blind participants to their allocated treatment regimen. Investigators are unable to package medications in a way other than that currently produced. It is the aim to outline, as part of the participant information and consent form (PICF), that both inhaled medications have proven to be efficacious (and detrimental in certain circumstances) in disease processes other than post lung transplant LRTI. Detection bias will be controlled by the use of a blinded outcome assessor for all follow-up data collection points.

Potential confounders in this study include the diagnosis of bronchiolitis obliterans (BOS), or chronic lung rejection, during which LRTI occurs simultaneously. Patients with a diagnosis of BOS may in fact demonstrate differences in lung physiology and ease of sputum expectoration, which may have an effect on outcomes variables. We feel that excluding these patients may have a detrimental impact on the external validity of this study, therefore we will stratify patients according to a diagnosis of BOS on study inclusion.

Outcomes and Significance This will be the first randomized controlled trial to analyze inhaled dornase alfa and isotonic saline in the post lung transplant population.

The outcome of this trial will help to guide physiotherapy and pharmacological management of post lung transplant patients with LRTI in the future, both nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Post bilateral sequential lung transplant
* Capable of performing airway clearance techniques / nebulisers
* Pulmonary exacerbation as defined by Fuchs et al
* Must be productive of sputum
* Able to provide informed consent within 48 hours of presentation.

  *Fuchs Scale(8): Treatment with / without parenteral antibiotics for 4/12 signs and symptoms:
* Change in sputum
* New or increased haemoptysis
* Increased cough
* Increased dyspnoea
* Malaise, fever or lethargy
* Temp above 38
* Anorexia or weight loss
* Sinus pain or tenderness
* Change in sinus discharge
* Change in physical examination of the chest
* Radiographic changes indicative of pulmonary infection
* Decrease in pulmonary function by 10 % or more

Exclusion Criteria:

* Paediatric transplant <18yrs
* Single lung transplant - native lung physiology may confound outcome measures
* Interstate - unable to complete follow up
* Unable to perform lung function testing
* Unable to complete subjective outcome measures- unable to read English fluently
* Critically unwell / intensive care unit / ventilator dependent
* Within 2 months of transplant date *Cystic Fibrosis will be stratified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Tarrant, B.Physio, Principal Investigator — The Alfred
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hertz MI. The Registry of the International Society for Heart and Lung Transplantation--Introduction to the 2012 annual reports: new leadership, same vision. J Heart Lung Transplant. 2012 Oct;31(10):1045-51. doi: 10.1016/j.healun.2012.08.003. No abstract available. PMID 22975094
- [Background] Herve P, Silbert D, Cerrina J, Simonneau G, Dartevelle P. Impairment of bronchial mucociliary clearance in long-term survivors of heart/lung and double-lung transplantation. The Paris-Sud Lung Transplant Group. Chest. 1993 Jan;103(1):59-63. doi: 10.1378/chest.103.1.59. PMID 8380268
- [Background] Munro PE, Button BM, Bailey M, Whitford H, Ellis SJ, Snell GI. Should lung transplant recipients routinely perform airway clearance techniques? A randomized trial. Respirology. 2008 Nov;13(7):1053-60. doi: 10.1111/j.1440-1843.2008.01386.x. Epub 2008 Aug 18. PMID 18721181
- [Background] Veale D, Glasper PN, Gascoigne A, Dark JH, Gibson GJ, Corris PA. Ciliary beat frequency in transplanted lungs. Thorax. 1993 Jun;48(6):629-31. doi: 10.1136/thx.48.6.629. PMID 8346493
- [Background] Humplik BI, Sandrock D, Aurisch R, Richter WS, Ewert R, Munz DL. Scintigraphic results in patients with lung transplants: a prospective comparative study. Nuklearmedizin. 2005 Apr;44(2):62-8. doi: 10.1267/nukl05020062. PMID 15861274
- [Background] Higenbottam T, Jackson M, Woolman P, Lowry R, Wallwork J. The cough response to ultrasonically nebulized distilled water in heart-lung transplantation patients. Am Rev Respir Dis. 1989 Jul;140(1):58-61. doi: 10.1164/ajrccm/140.1.58. PMID 2502056
- [Background] Fuchs HJ, Borowitz DS, Christiansen DH, Morris EM, Nash ML, Ramsey BW, Rosenstein BJ, Smith AL, Wohl ME. Effect of aerosolized recombinant human DNase on exacerbations of respiratory symptoms and on pulmonary function in patients with cystic fibrosis. The Pulmozyme Study Group. N Engl J Med. 1994 Sep 8;331(10):637-42. doi: 10.1056/NEJM199409083311003. PMID 7503821
- [Background] Touleimat BA, Conoscenti CS, Fine JM. Recombinant human DNase in management of lobar atelectasis due to retained secretions. Thorax. 1995 Dec;50(12):1319-21; discussion 1323. doi: 10.1136/thx.50.12.1319. PMID 8553310
- [Background] Voelker KG, Chetty KG, Mahutte CK. Resolution of recurrent atelectasis in spinal cord injury patients with administration of recombinant human DNase. Intensive Care Med. 1996 Jun;22(6):582-4. doi: 10.1007/BF01708100. PMID 8814475
- [Background] Riethmueller J, Borth-Bruhns T, Kumpf M, Vonthein R, Wiskirchen J, Stern M, Hofbeck M, Baden W. Recombinant human deoxyribonuclease shortens ventilation time in young, mechanically ventilated children. Pediatr Pulmonol. 2006 Jan;41(1):61-6. doi: 10.1002/ppul.20298. PMID 16265663
- [Background] Crockett AJ, Cranston JM, Latimer KM, Alpers JH. Mucolytics for bronchiectasis. Cochrane Database Syst Rev. 2000;(2):CD001289. doi: 10.1002/14651858.CD001289. PMID 10796636
- [Background] Wark P, McDonald VM. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD001506. doi: 10.1002/14651858.CD001506.pub3. PMID 19370568
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Nicolson CH, Stirling RG, Borg BM, Button BM, Wilson JW, Holland AE. The long term effect of inhaled hypertonic saline 6% in non-cystic fibrosis bronchiectasis. Respir Med. 2012 May;106(5):661-7. doi: 10.1016/j.rmed.2011.12.021. Epub 2012 Feb 19. PMID 22349069
- [Background] Safdar A, Shelburne SA, Evans SE, Dickey BF. Inhaled therapeutics for prevention and treatment of pneumonia. Expert Opin Drug Saf. 2009 Jul;8(4):435-49. doi: 10.1517/14740330903036083. PMID 19538104
- [Background] Amin R, Subbarao P, Lou W, Jabar A, Balkovec S, Jensen R, Kerrigan S, Gustafsson P, Ratjen F. The effect of dornase alfa on ventilation inhomogeneity in patients with cystic fibrosis. Eur Respir J. 2011 Apr;37(4):806-12. doi: 10.1183/09031936.00072510. Epub 2010 Aug 6. PMID 20693248
- [Background] Amin R, Subbarao P, Jabar A, Balkovec S, Jensen R, Kerrigan S, Gustafsson P, Ratjen F. Hypertonic saline improves the LCI in paediatric patients with CF with normal lung function. Thorax. 2010 May;65(5):379-83. doi: 10.1136/thx.2009.125831. PMID 20435858
- [Background] Raj AA, Pavord DI, Birring SS. Clinical cough IV:what is the minimal important difference for the Leicester Cough Questionnaire? Handb Exp Pharmacol. 2009;(187):311-20. doi: 10.1007/978-3-540-79842-2_16. PMID 18825348
- [Background] Jones PW. Interpreting thresholds for a clinically significant change in health status in asthma and COPD. Eur Respir J. 2002 Mar;19(3):398-404. doi: 10.1183/09031936.02.00063702. PMID 11936514
- [Background] Leidy NK, Rennard SI, Schmier J, Jones MK, Goldman M. The breathlessness, cough, and sputum scale: the development of empirically based guidelines for interpretation. Chest. 2003 Dec;124(6):2182-91. doi: 10.1378/chest.124.6.2182. PMID 14665499
- [Background] Stockley RA, Bayley D, Hill SL, Hill AT, Crooks S, Campbell EJ. Assessment of airway neutrophils by sputum colour: correlation with airways inflammation. Thorax. 2001 May;56(5):366-72. doi: 10.1136/thorax.56.5.366. PMID 11312405

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dornase Alfa | Isotonic Saline
Started | 16 | 16
ITT Analysis | 16 | 16
Discontinued Intervention | 2 | 1
Death | 1 | 1
Missing Baseline LCI 2% Data. | 0 | 2
Missing 1+3 Month LCI 2% Data. | 2 | 1
Missing 3 Month LCI 2% Data. | 1 | 0
Completed (Complete data for primary outcome.) | 13 | 13
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Dornase Alfa: Once daily, 2.5ml inhaled dornase alfa.
  Dornase Alfa: Once daily, 2.5ml inhaled dornase alpha (evening if able) with inhalational breathing routine (IBR). IBR consists of 4 slow deep breaths followed by 6 relaxed breaths, repeated until nebuliser is complete, coughing when the patient feels the need to expectorate. The patient will be instructed to sit in an upright position with upper limb support as able.
- Total: Total of all reporting groups
Arm/Group | Dornase Alfa | Isotonic Saline | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.88 (10.77) | 47.56 (15.99) | 50.22 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 11 | 7 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 16 | 16 | 32
Days since transplant [Median (Inter-Quartile Range); unit: Days] | 1162.50 [127.75 to 2559.25] | 1497 [194.75 to 3014.50] | 1275 [146.50 to 2628.25]
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 24.94 (4.95) | 23.96 (6.10) | 24.45 (5.48)
Chronic Lung Allograft Dysfunction (CLAD) diagnosis at baseline [Count of Participants; unit: Participants] | 2 | 5 | 7
Sinus disease diagnosis at baseline [Count of Participants; unit: Participants] | 4 | 2 | 6
Gastro-Oesophageal Reflux Disease (GORD) diagnosis at baseline [Count of Participants; unit: Participants] | 12 | 13 | 25
Initial inpatient length of stay (LOS) [Median (Inter-Quartile Range); unit: Days] | 6.5 [4.25 to 9.50] | 7.0 [5.50 to 9.75] | 7.0 [5.0 to 9.75]
C-Reactive Protein (CRP) [Median (Inter-Quartile Range); unit: mg/L] | 6 [1.00 to 30.50] | 29.50 [2.00 to 75.75] | 9.00 [1.00 to 45.00]
Multiple Breath Washout (MBW) [Mean (Standard Deviation); unit: Index] — Multiple breath washout is a sensitive measure of respiratory function performed with the subject in a seated position, breathing a fixed tidal volume (1L) of inert gas (nitrogen) from functional residual capacity (FRC) via mouthpiece.
  Two common outcomes of MBW are Sacin, a measure of gas mixing at the diffusion front, or acinar entrance in the airways, and Scond, in the proximal, conductive zones. An increase in either Sacin or Scond represents an increase in ventilation heterogeneity (deterioration). Both increase with age, normal values are non-zero between 0-0.25(Sacin) and 0-0.1(Scond). Population: Baseline MBW data lost due to technical error (IS n=2)
  Index
    Sacin: number analyzed (Participants) | 16 | 14 | 30
    Sacin | 0.337 (0.173) | 0.354 (0.218) | 0.345 (0.191)
    Scond: number analyzed (Participants) | 16 | 14 | 30
    Scond | 0.035 (0.026) | 0.026 (0.023) | 0.031 (0.025)
Lung Clearance Index (2%) [Mean (Standard Deviation); unit: Index] — Amount of lung volume turnovers required to clear nitrogen to 2% of starting concentration. Population: Baseline data lost due to technical error (Isotonic saline (IS) group n=2)
  Index
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 10.31 (2.38) | 11.05 (2.40) | 10.65 (2.38)
Forced Expiratory Ratio (FER) [Mean (Standard Deviation); unit: Ratio] | 61.56 (13.28) | 69.31 (12.05) | 65.44 (13.08)
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Liters (L)] | 1.95 (0.77) | 1.65 (0.74) | 1.80 (0.76)
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Percent (%)] | 62.50 (25.11) | 53.00 (18.55) | 57.75 (22.25)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Liters (L)] | 3.10 (0.84) | 2.36 (0.85) | 2.73 (0.91)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Percent (%)] | 75.18 (19.29) | 59.81 (14.07) | 67.81 (18.49)
Functional Residual Capacity [Mean (Standard Deviation); unit: Liters (L)] — Population: Baseline data lost due to technical error (Isotonic saline (IS) group n=2)
  Liters (L)
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 2.32 (0.86) | 1.83 (0.76) | 2.09 (0.84)
Leicester Cough Questionnaire (LCQ) [Mean (Standard Deviation); unit: units on a scale] — Cough specific quality of life (QOL). Scale 1-7 for physical, psychological, social. Scale 3-21 for total. Lower=worse.
  units on a scale
    Physical | 4.53 (1.04) | 4.69 (1.17) | 4.61 (1.09)
    Psychological | 4.68 (1.35) | 4.95 (1.69) | 4.81 (1.51)
    Social | 4.98 (1.57) | 4.95 (1.62) | 4.97 (1.57)
    Total | 14.44 (3.88) | 14.60 (4.25) | 14.52 (4.00)
St George's Respiratory Questionnaire (SGRQ) [Mean (Standard Deviation); unit: units on a scale] — Respiratory specific QOL. 50 items, 76 weighted responses. Scores range 0-100, higher=worse.
  units on a scale
    Symptom | 55.51 (19.59) | 53.35 (16.92) | 54.43 (18.04)
    Activity | 50.37 (29.25) | 58.25 (21.34) | 54.31 (25.50)
    Impact | 30.53 (17.61) | 34.06 (14.39) | 32.30 (15.92)
    Total | 40.64 (19.78) | 44.69 (14.82) | 42.66 (17.32)

OUTCOME MEASURES:

1. Primary Outcome: Lung Clearance Index 2% (LCI2%)
Description: A measure of ventilation inhomogeneity as measured during multiple breath washout (MBW) of inert tracer gases. It has been shown that this test is a potentially more sensitive measure of peripheral airway obstruction than regular spirometry in short term (4 week) mucolytic interventional studies in pediatric Cystic Fibrosis (CF)(17-18). This test would be performed within the respiratory physiology lung function laboratory on site at all assessment points, by an assessor who is blinded to group allocation for follow up data collection.
  Conventionally used primary endpoints in this population, such as regular spirometry(3), may be unable to detect between group differences without large sample sizes and long treatment durations. Based on current evidence from non-lung transplant populations, LCI has been able to show short-term change, whereas regular spirometry has not shown change(17-18).
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Index (change)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 14 | 15
Index (change)
  1 month | 10.68 (1.97) | 11.65 (2.33)
  3 months: number analyzed (Participants) | 13 | 15
  3 months | 10.09 (2.19) | 11.19 (2.73)

2. Secondary Outcome: Multiple Breath Washout (MBW)
Description: Multiple breath washout is a sensitive measure of respiratory function performed with the subject in a seated position, breathing a fixed tidal volume (1L) of inert gas (nitrogen) from functional residual capacity (FRC) via mouthpiece.
  Two common outcomes of MBW are Sacin, a measure of gas mixing at the diffusion front, or acinar entrance in the airways, and Scond, in the proximal, conductive zones. An increase in either Sacin or Scond represents an increase in ventilation heterogeneity (deterioration). Both increase with age, normal values are non-zero between 0-0.25(Sacin) and 0-0.1(Scond).
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Gas mixing index (Sacin / Scond)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 14 | 15
Gas mixing index (Sacin / Scond)
  Sacin 1 month | 0.348 (0.155) | 0.383 (0.227)
  Sacin 3 months: number analyzed (Participants) | 13 | 15
  Sacin 3 months | 0.354 (0.249) | 0.356 (0.188)
  Scond 1 month | 0.045 (0.037) | 0.026 (0.037)
  Scond 3 months: number analyzed (Participants) | 13 | 15
  Scond 3 months | 0.033 (0.017) | 0.021 (0.027)

3. Secondary Outcome: Functional Residual Capacity (FRC)
Description: Volume of air remaining in the lungs after normal expiration.
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 14 | 15
Liters (L)
  1 month | 2.03 (0.96) | 1.80 (0.81)
  3 months: number analyzed (Participants) | 13 | 15
  3 months | 2.22 (1.01) | 1.78 (0.76)

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Liters
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: 1 month, 3 months.
Population: Dropout
Measure: Mean (Standard Deviation); unit: Liters (L) - change
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 15 | 15
Liters (L) - change
  FEV1 L 1 month | 2.11 (0.68) | 1.76 (0.81)
  FEV1 L 3 months: number analyzed (Participants) | 14 | 15
  FEV1 L 3 months | 1.91 (0.88) | 1.78 (0.82)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Percent.
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 15 | 15
Percent (%)
  1 month | 69.33 (25.35) | 58.33 (21.44)
  3 months: number analyzed (Participants) | 14 | 15
  3 months | 63.00 (27.94) | 57.60 (22.35)

6. Secondary Outcome: Forced Vital Capacity (FVC) Liters
Description: Forced vital Capacity (FVC) is a measure of the amount of air someone can forcibly expel out of the lungs after taking a breath to fill the lungs as much as possible.
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 15 | 15
Liters (L)
  1 month | 3.21 (0.73) | 2.46 (0.91)
  3 months: number analyzed (Participants) | 14 | 15
  3 months | 2.96 (0.75) | 2.50 (0.89)

7. Secondary Outcome: Forced Vital Capacity (FVC) Percent
Description: as for outcome 6
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 15 | 15
Percent (%)
  1 month | 79.40 (18.07) | 62.07 (16.34)
  3 months: number analyzed (Participants) | 14 | 15
  3 months | 74.41 (17.02) | 63.73 (16.88)

8. Secondary Outcome: Forced Expiratory Ratio (FER)
Description: FER represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
Time Frame: 1 month, 3 months
Population: Dropout
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 15 | 15
Ratio
  1 month | 66.33 (14.03) | 70.87 (11.95)
  3 months: number analyzed (Participants) | 14 | 15
  3 months | 62.79 (17.13) | 70.27 (13.67)

9. Secondary Outcome: Leicester Cough Questionnaire (LCQ) - Change
Description: Cough specific quality of life questionnaire. The LCQ is a 19-question tool, validated in chronic lung disease other than lung transplant(19). Scale 1-7 for physical, psychological, social. Combined score of 3-21 for total. Lower=worse.
Time Frame: 1 month, 3 months.
Population: Dropout / loss of data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 15
score on a scale
  Physical 1 month: number analyzed (Participants) | 16 | 13
  Physical 1 month | 5.73 (0.86) | 5.12 (0.90)
  Physical 3 months: number analyzed (Participants) | 15 | 15
  Physical 3 months | 5.56 (1.25) | 5.69 (0.89)
  Psychological 1 month: number analyzed (Participants) | 16 | 13
  Psychological 1 month | 6.32 (0.87) | 5.87 (0.96)
  Psychological 3 months: number analyzed (Participants) | 15 | 15
  Psychological 3 months | 6.03 (1.35) | 6.05 (0.95)
  Social 1 month: number analyzed (Participants) | 16 | 13
  Social 1 month | 6.33 (0.77) | 5.75 (0.97)
  Social 3 months: number analyzed (Participants) | 15 | 15
  Social 3 months | 6.12 (1.18) | 6.07 (0.98)
  Total 1 month: number analyzed (Participants) | 16 | 13
  Total 1 month | 17.26 (4.62) | 16.72 (2.51)
  Total 3 months: number analyzed (Participants) | 15 | 15
  Total 3 months | 17.70 (3.69) | 17.81 (2.71)

10. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) - Change
Description: The SGRQ is a 2-part questionnaire, validated in chronic lung disease other than lung transplant(20).
  50 items, 76 weighted responses. Scores range 0-100, higher=worse.
Time Frame: 1 month, 3 months.
Population: Dropout / lost data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 15
units on a scale
  Symptom 1 month: number analyzed (Participants) | 16 | 13
  Symptom 1 month | 55.65 (19.25) | 61.93 (17.45)
  Symptom 3 months: number analyzed (Participants) | 15 | 14
  Symptom 3 months | 48.52 (17.54) | 51.47 (23.03)
  Activity 1 month: number analyzed (Participants) | 16 | 13
  Activity 1 month | 40.82 (25.31) | 57.38 (22.59)
  Activity 3 months: number analyzed (Participants) | 15 | 15
  Activity 3 months | 53.18 (32.15) | 53.81 (29.58)
  Impact 1 month: number analyzed (Participants) | 16 | 13
  Impact 1 month | 20.59 (17.47) | 30.72 (13.49)
  Impact 3 months: number analyzed (Participants) | 15 | 15
  Impact 3 months | 25.96 (21.54) | 33.90 (22.16)
  Total 1 month: number analyzed (Participants) | 16 | 13
  Total 1 month | 32.50 (17.98) | 43.58 (14.28)
  Total 3 months: number analyzed (Participants) | 15 | 14
  Total 3 months | 37.97 (22.75) | 40.81 (22.63)

11. Secondary Outcome: Inpatient Days
Description: Number of days spent in the acute inpatient setting.
Time Frame: Across study period (3 months).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 16
Days
  All cause - intervention | 8.67 (3.88) | 12.50 (15.76)
  All cause - follow-up | 8.09 (7.73) | 11.38 (10.07)
  Respiratory - intervention | 9.20 (4.09) | 21.50 (20.51)
  Respiratory - follow-up | 9.83 (9.24) | 14.33 (9.99)

12. Secondary Outcome: Oral, Inhaled or Intravenous Antibiotic (IVAB) Days.
Description: Antibiotic use for the treatment of lower respiratory tract infections (LRTI) only.
Time Frame: Over study period (3 months).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 16
Days
  Intervention phase | 23.50 [14.00 to 30.00] | 25.00 [17.50 to 29.75]
  Follow-up phase | 14.00 [0 to 32.25] | 10.50 [0 to 34.50]

13. Secondary Outcome: Number of Hospitalizations
Description: Number of admissions to the acute setting.
Time Frame: Over study period (3 months).
Measure: Number; unit: Hospitalizations
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 16
Hospitalizations
  All cause - intervention | 8 | 4
  All cause - follow-up | 12 | 8
  Respiratory - intervention | 7 | 2
  Respiratory - follow-up | 6 | 6

14. Secondary Outcome: C-reactive Protein (CRP)
Description: An inflammatory marker measured with routine blood tests on admission with LRTI. Taken during inpatient (IP) stay and routinely on outpatient (OP) follow-up. Existing / available data only will be used - no extra routine bloods will be taken on account of study inclusion.
Time Frame: 1 month, 3 months.
Population: Data only available when routinely collected.
Measure: Median (Inter-Quartile Range); unit: mg/L (change)
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 10 | 10
mg/L (change)
  1 month | 1.00 [1.00 to 9.25] | 2.50 [1.00 to 32.00]
  3 months: number analyzed (Participants) | 7 | 10
  3 months | 12 [1.00 to 24.00] | 1.00 [1.00 to 70.50]

15. Secondary Outcome: Breathlessness, Cough and Sputum Scale (BCSS) - Exacerbations
Description: Self-reported symptom severity, used as a daily patient diary. The BCSS is a 12 point self-reported symptom severity score, consisting of 3 sections concerning how much difficulty the subject is having with breathing; subjective cough symptoms and trouble caused by sputum, each scoring between 0-4, combining to a total score of 0-12 (higher=worse). This scale is validated for daily use in Chronic Obstructive Pulmonary Disease (COPD)(21).
  An exacerbation was defined as an increase in BCSS>1 with ≥5 days preceding stability.
Time Frame: Daily up to 3 months.
Measure: Mean (Standard Deviation); unit: Exacerbations
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 16
Exacerbations
  Intervention phase | 0.94 (1.00) | 1.07 (1.00)
  Follow-up phase | 2.64 (2.02) | 3.62 (2.02)

16. Secondary Outcome: BronkoTest (Sputum Colour) - Purulent Sputum Days
Description: Sputum colour chart. Sputum colour has been shown to correlate with physiological infection in other chronic lung disease groups(22).
Time Frame: Daily up to 3 months.
Population: Dropout / loss of data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dornase Alfa | Isotonic Saline
Number analyzed (Participants) | 16 | 14
days
  Intervention phase | 11.50 [5.50 to 22.50] | 8.50 [4.00 to 18.25]
  Follow-up phase: number analyzed (Participants) | 14 | 13
  Follow-up phase | 4.50 [0 to 22.50] | 6.00 [1.50 to 15.00]

ADVERSE EVENTS:
Time Frame: Adverse events: Baseline to 1 month. Mortality: Baseline to 3 months.
Description: Adverse events specifically related to intervention administration were collected by way of medial record review as inpatient, and/or patient diary as an outpatient. Adverse events were screened for daily whilst an inpatient, and at the first scheduled follow up assessment as an outpatient at the point cessation of intervention (1 month).
  All-cause mortality was recorded across the entire study period (Baseline to 3 months).
Arm/Group | Dornase Alfa | Isotonic Saline
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dornase Alfa (N=16) | Isotonic Saline (N=16)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pre-existing/new diagnoses CLAD +/- LRTI; Participants deviating from protocol; Potential for performance bias; Infection control excluded viral LRTI; Single center trial; Participants were >2 months post-tx.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT01952470/Prot_SAP_000.pdf
  • Informed Consent Form (2014-09-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT01952470/ICF_001.pdf